CLINICAL TRIAL: NCT00594919
Title: Neutrophil Gelatinase-Associated Lipocalin(NGAL): Early Biomarker of Acute Kidney Injury After Cardiac Surgery
Brief Title: Neutrophil Gelatinase-Associated Lipocalin: Biomarker of Acute Kidney Injury After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Base (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Fundação de Amparo à Pesquisa do Estado de São Paulo, FAPESP
Other Study IDs: CAAE 0246.0.000.140-07; 1411 - 2007.
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Early Acute Kidney Injury
Keywords: acute kidney injury; ngal; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AKI group: Acute kidney injury group after cardiac surgery.
- NKF group: Normal kidney function group after cardiac surgery

SUMMARY:
The following objectives were used for comparison: 1)primary objective: Evaluate the urinary excretion of NGAL as a marker of early development of acute kidney injury in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
All patients aged greater than 18 years undergoing elective cardiac surgery for coronary artery bypass grafting and / or valve replacement, in need of cardiopulmonary bypass and with the prospect of minimum hospital length stay of 48 hours in ICU, will be candidates for participation in this study.

Criteria for exclusion Patients with IRA before hospitalization in the ICU; Patients with estimated glomerular filtration (MDRD formula simplified) less than 30 ml / min; Patients transplanted kidney; Patients with chronic renal failure on dialysis; Patients anuric the admission in the ICU; Refusal to participate in the study.

Definition of IRA:

IRA will be defined according to the new proposal of AKIN (Acute Kidney Injury Network) (awaiting publication): abrupt elevation (48 hours) of serum creatinine in value greater than or equal to 0.3 mg / dL or an increase of 50% compared to baseline or reduction of urinary volume to 0.5 ml / kg / h for more than 6 hours (Annex 1).

Laboratory Investigations Samples of urine will be collected before surgery, after 2, 4, 6, 12, 24, 48, 72 and 96 hours after the end of the CEC for determination of creatinine and urinary NGAL (normalization of NGAL for excretion urinary creatinine).

The serum creatinine is measured before surgery and daily during the first 4 days after surgery for the diagnosis of IRA. If the time of CEC exceed 2 hours, the first sample of urine after the end of the CEC will be considered as "sample 2 hours".

Quantification of NGAL Samples of urine will be centrifuged (5 min at 2000 rpm) and frozen at -20 ° C for later determination of NGAL by method of ELISA (Kit commercial AntybodyShop, Denmark).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than 18 years undergoing elective cardiac surgery for coronary artery bypass grafting and/or valve replacement
* In need of cardiopulmonary bypass and with the prospect of minimum hospital length stay of 48 hours in ICU

Exclusion Criteria:

* Patients with IRA before hospitalization in the ICU
* Patients with estimated glomerular filtration (MDRD formula simplified) less than 30 ml/min
* Patients transplanted kidney
* Patients with chronic renal failure on dialysis
* Patients anuric the admission in the ICU
* Refusal to participate in the study.

Definition of IRA:

IRA will be defined according to the new proposal of AKIN (Acute Kidney Injury Network) (awaiting publication): abrupt elevation (48 hours) of serum creatinine in value greater than or equal to 0.3 mg / dL or an increase of 50% compared to baseline or reduction of urinary volume to 0.5 ml / kg / h for more than 6 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged greater than 18 years undergoing elective cardiac surgery for coronary artery bypass grafting and / or valve replacement, in need of cardiopulmonary bypass and with the prospect of minimum hospital length stay of 48 hours in ICU, will be candidates for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Evaluate the urinary excretion of NGAL as a marker of early development of acute kidney injury in patients undergoing cardiac surgery | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Emerson quintino, Study Director — Hospital de Base
Locations (1):
- Hospital de Base - São José do Rio preto Medical School, São José do Rio Preto, São Paulo, Brazil